CLINICAL TRIAL: NCT03109873
Title: Pilot Study of Metformin in Head and Neck Cancer and Its Effect on Proinflammatory Cytokines and Exosomes Implicated in Acute and Chronic Toxicity
Brief Title: Metformin Hydrochloride in Affecting Cytokines and Exosomes in Patients With Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16D.639; JT 9410 (Other: JeffTrial Number)
Record Dates: First submitted 2017-03-06; First posted 2017-04-12 (Actual); Results first posted 2019-11-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Larynx; Lip; Oral Cavity; Pharynx
MeSH Terms: conditions — Laryngeal Diseases; Lymphoid Interstitial Pneumonia | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (EBRT, metformin hydrochloride) (Experimental): Patients undergo External Beam Radiation Therapy (EBRT). Beginning 1 week prior to start of EBRT, patients receive metformin hydrochloride PO QD for 3 days and BID thereafter until 2 weeks after completion of EBRT.
  Interventions: Radiation: External Beam Radiation Therapy; Drug: Metformin Hydrochloride
- Arm II (EBRT, placebo) (Placebo Comparator): Patients undergo External Beam Radiation Therapy (EBRT). Beginning 1 week prior to start of EBRT, patients receive placebo PO QD for 3 days and BID thereafter until 2 weeks after completion of EBRT.
  Interventions: Radiation: External Beam Radiation Therapy; Other: Placebo

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo External Beam Radiation Therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam RT
Drug: Metformin Hydrochloride — Given orally
  Other Names: 1,1-Dimethylbiguanide Hydrochloride; 1115-70-4; 91485; Cidophage; Glucoformin; Glucophage ER; Dimefor
  Arms: Arm I (EBRT, metformin hydrochloride)
Other: Placebo — Given orally
  Arms: Arm II (EBRT, placebo)

SUMMARY:
This pilot clinical trial studies how well metformin hydrochloride works in affecting cytokines and exosomes in patients with head and neck cancer. Metformin hydrochloride may reduce the metabolic activity of cancer cells and of surrounding supportive tissues.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the capacity of metformin hydrochloride (metformin) to alter the cytokine and exosome profiles.

II. To assess the capacity of metformin to mitigate known side effects of external beam radiation therapy including inflammation, mucositis, dysphagia, xerostomia, and fatigue.

SECONDARY OBJECTIVES:

I. Assess safety and tolerability of metformin treatment in subjects undergoing external beam radiation treatment for head and neck cancer.

II. To determine the effect of metformin treatment on symptoms of xerostomia as assessed by the Xerostomia Questionnaire (XQ).

III. To determine the effect of metformin treatment on symptoms of mucositis as assessed by World Health Organization (WHO) classification.

IV. To determine the effect of metformin treatment on symptoms of dysphagia as assessed by the MD Anderson Dysphagia Inventory.

V. To determine the effect of metformin treatment on symptoms of fatigue as assess by the Multidimensional Fatigue Inventory (MFI).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of head and neck cancer biopsy proven, and who are candidates for radiation therapy
* All subjects must be able to comprehend and sign a written informed consent document.

Exclusion Criteria:

* Subjects who are pregnant or may become pregnant during metformin administration; pregnancy testing will be done in conjunction with preradiation protocols
* Subjects on metformin for any reason during the preceding 4 weeks
* Diabetic subjects are eligible if they are not taking metformin or insulin
* Subjects who have received iodinated contrast dye must wait 12 hours prior to starting Metformin. If a CT scan with contrast is scheduled after screening and consent, the metformin cannot be taken until after the CT with contrast has been completed and they have waited 12 hours.
* Patients with plasma creatinine level greater than 1.3 mg/dL
* Patients with plasma bicarbonate less than 22 mEq/L or history of lactic or any other metabolic acidosis
* Patients with history of congestive heart failure
* Patients with myocardial ischemia or peripheral muscle ischemia
* Patients with sepsis or severe infection
* Patients with history of lung disease currently requiring any supplemental oxygen treatment
* Patients scheduled for radiation less than 6 days from enrollment
* Patients with history of hepatic dysfunction or hepatic disease and abnormal liver function tests; patients who have a history of hepatic dysfunction or hepatic disease and normal liver function tests will be eligible to participate
* Patients with a current history (in the past 30 days) of heaving drinking which is defined in accordance with CDC definition as more than 8 drinks per week for women and more than 15 drinks per week for men. A standard drink contains .6 ounces of pure alcohol. Generally, this amount of pure alcohol is found in 12-ounces of beer, 8-ounces of malt liquor, 5-ounces of wine, 1.5-ounces or a "shot" of 80-proof distilled spirits or liquor (e.g., gin, rum, vodka, or whiskey). While on study, patients should limit their alcohol consumption to no more than 8 drinks per week for women and no more than 15 drinks per week for men. Patients who feel they cannot comply with this recommendation are not eligible".
* All medications are permitted except those that are contraindicated with metformin under current Food and Drug Administration (FDA) recommendations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Luginbuhl, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (EBRT, Metformin Hydrochloride) | Arm II (EBRT, Placebo)
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (EBRT, Metformin Hydrochloride) | Arm II (EBRT, Placebo) | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cytokine/Chemokine Profile
Description: Mixed effects linear regression will be used to model longitudinal measurements of each cytokine.
Time Frame: Up to 1 year
Population: Due to insufficient accrual, statistical results cannot be reported.
Arm/Group | Arm I (EBRT, Metformin Hydrochloride) | Arm II (EBRT, Placebo)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mucositis Assessed Using WHO Classification
Description: Analysis will be primarily descriptive. The distribution of swallowing function and mucositis scores will be summarized by arm using means, medians, standard deviations, and ranges.
Time Frame: Up to 1 year
Population: Due to insufficient accrual, statistical results cannot be reported.
Arm/Group | Arm I (EBRT, Metformin Hydrochloride) | Arm II (EBRT, Placebo)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Objective Response Rate
Description: The objective response rate will be estimated by arm along with an exact 95% binomial confidence interval
Time Frame: Up to 2 years
Population: Due to insufficient accrual, statistical results cannot be reported.
Arm/Group | Arm I (EBRT, Metformin Hydrochloride) | Arm II (EBRT, Placebo)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Exosome Profile
Description: Longitudinal measurements of exosomes will also be modeled using mixed effects linear regression. This analysis is treated as separate from the cytokine questions and the p-value will not be adjusted.
Time Frame: Up to 1 year
Population: Due to insufficient accrual, statistical results cannot be reported.
Arm/Group | Arm I (EBRT, Metformin Hydrochloride) | Arm II (EBRT, Placebo)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Toxicities
Description: Evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to 2 years
Population: Due to insufficient accrual, statistical results cannot be reported.
Arm/Group | Arm I (EBRT, Metformin Hydrochloride) | Arm II (EBRT, Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: baseline through one year after completion of treatment
Arm/Group | Arm I (EBRT, Metformin Hydrochloride) | Arm II (EBRT, Placebo)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 4/5 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (EBRT, Metformin Hydrochloride) (N=5) | Arm II (EBRT, Placebo) (N=4)
Xerostomia (General disorders) | 4 | 2 — Dry mouth
Dysphagia (General disorders) | 4 | 2
Fatigue (General disorders) | 4 | 3
Dysgeusia (General disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT03109873/Prot_SAP_000.pdf